CLINICAL TRIAL: NCT00452452
Title: A Phase 3 Open-label Trial Evaluating the Safety, Tolerability and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Older Infants and Children Who Are Naive to Previous Vaccination With Pneumococcal Conjugate Vaccine.
Brief Title: Study Evaluating 13-valent Pneumococcal Conjugate Vaccine Catch-Up Regimens in Older Infants and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6096A1-3002
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Results first posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-07

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal Vaccines
MeSH Terms: conditions — Pneumococcal Infections

ARMS (1):
- A (Experimental)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent Pneumococcal conjugate vaccine (13vPnC) in older infants and children who have not previously been immunized with Pneumococcal vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 7 months to <72 months at time of enrollment.
2. Available for entire study period and whose parent/legal guardian could be reached by telephone.
3. Healthy as determined by medical history, physical examination, and judgment of the investigator.
4. Parent/legal guardian had to be able to complete all relevant study procedures during subject participation.

Exclusion Criteria:

1. Previous vaccination with licensed or investigational pneumococcal vaccine.
2. A previous anaphylactic reaction to any vaccine or vaccine-related component.
3. Contraindication to vaccination with pneumococcal vaccine.
4. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
5. Known or suspected immune deficiency or suppression.
6. History of culture-proven invasive disease caused by S pneumoniae.
7. Major known congenital malformation or serious chronic disorders.
8. Significant neurological disorder or history of seizure including febrile seizure, or significant stable or evolving disorders such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorders. Does not include resolving syndromes due to birth trauma such as Erb palsy.
9. Receipt of blood products or gamma-globulin (including monoclonal antibodies) in the last 3 months.
10. Participation in another investigational or interventional trial. Participation in purely observational studies is acceptable.
11. Child is a direct descendant (child or grandchild) of a member of the study site personnel.

Ages: 7 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 355 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Poland: WPWZMED@wyeth.com
Locations (8):
- Poland (8):
  - Bydgoszcz
  - Dębica
  - Krakow
  - Lodz
  - Oborniki Salskie
  - Proznan
  - Trzebnica
  - Łęczna

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Poland from July 2007 to September 2007.
Pre-assignment Details: Participants were enrolled into the study according to inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC 7 to <12 Months of Age: Participants 7 to less than (<) 12 months of age with 0 prior doses of 7-valent pneumococcal conjugate vaccine (Prevnar) received a total of 3 single intramuscular (IM) 0.5 milliliter (mL) doses of 13-valent pneumococcal conjugate vaccine (13vPnC); the first two at least 28 days apart (infant series) and the third single IM 0.5 mL dose of 13vPnC at 12 to 16 months of age (toddler dose), at least 46 days after last infant dose.
- 13vPnC 12 to <24 Months of Age: Participants 12 to < 24 months of age with 0 prior dose of 7-valent pneumococcal conjugate vaccine (Prevnar) received a total of 2 single IM 0.5 mL doses of 13vPnC at least 56 days apart.
- 13vPnC 24 to < 72 Months of Age: Participants 24 to < 72 months of age with 0 prior doses of 7-valent pneumococcal conjugate vaccine (Prevnar) received a single IM 0.5 mL dose of 13vPnC.
Period: Overall Study
Arm/Group | 13vPnC 7 to <12 Months of Age | 13vPnC 12 to <24 Months of Age | 13vPnC 24 to < 72 Months of Age
Started | 90 | 112 | 153
Vaccinated Dose 1 | 90 | 112 | 152
Vaccinated Dose 2 | 90 | 112 | 0
Vaccinated Dose 3 | 89 | 0 | 0
Completed | 88 | 112 | 152
Not Completed | 2 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC 7 to <12 Months of Age | 13vPnC 12 to <24 Months of Age | 13vPnC 24 to < 72 Months of Age | Total
Number analyzed (Participants) | 90 | 112 | 153 | 355
Age Continuous [Mean (Standard Deviation); unit: months] | 8.7 (1.6) | 17.6 (3.5) | 42.0 (13.1) | 25.9 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 58 | 74 | 179
  Male | 43 | 54 | 79 | 176

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Antibody Level ≥0.35μg/mL After Vaccination
Description: Percentages of participants achieving World Health Organization (WHO) predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: 28 to 42 days after vaccination 3 for Group 1 (13 to <17 months of age), after vaccination 2 for Group 2 (14 to <26 months of age), and after vaccination 1 for Group 3 (26 to <73 months of age).
Population: Evaluable immunogenicity (per protocol) population who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate immunoglobulin G (IgG) antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC 7 to <12 Months of Age | 13vPnC 12 to <24 Months of Age | 13vPnC 24 to < 72 Months of Age
Number analyzed (Participants) | 84 | 110 | 152
percentage of participants
  Common Serotypes - Serotype 4 (n= 84,110,151) | 100.0 [95.7 to 100.0] | 100.0 [96.7 to 100.0] | 99.3 [96.4 to 100.0]
  Common Serotypes - Serotype 6B (n=83,110,150) | 98.8 [93.5 to 100.0] | 100.0 [96.7 to 100.0] | 99.3 [96.3 to 100.0]
  Common Serotypes - Serotype 9V (n= 83,104,148) | 98.8 [93.5 to 100.0] | 99.0 [94.8 to 100.0] | 98.6 [95.2 to 99.8]
  Common Serotypes - Serotype 14 (n= 84,108,135) | 100.0 [95.7 to 100.0] | 100.0 [96.6 to 100.0] | 88.1 [81.5 to 93.1]
  Common Serotypes - Serotype 18C (n= 83,109,151) | 100.0 [95.7 to 100.0] | 100.0 [96.7 to 100.0] | 98.7 [95.3 to 99.8]
  Common Serotypes - Serotype 19F (n=84,110,147) | 97.6 [91.7 to 99.7] | 100.0 [96.7 to 100.0] | 98.0 [94.2 to 99.6]
  Common Serotypes - Serotype 23F (n= 84,110,151) | 98.8 [93.5 to 100.0] | 92.7 [86.2 to 96.8] | 93.4 [88.2 to 96.8]
  Additional Serotypes - Serotype 1 (n= 83,108,149) | 100.0 [95.7 to 100.0] | 100.0 [96.6 to 100.0] | 96.6 [92.3 to 98.9]
  Additional Serotypes - Serotype 3 (n= 83,108,149) | 98.8 [93.5 to 100.0] | 100.0 [96.6 to 100.0] | 97.3 [93.3 to 99.3]
  Additional Serotypes - Serotype 5 (n= 84,107,152) | 97.6 [91.7 to 99.7] | 99.1 [94.9 to 100.0] | 98.7 [95.3 to 99.8]
  Additional Serotypes - Serotype 6A (n= 84,110,150) | 100.0 [95.7 to 100.0] | 98.2 [93.6 to 99.8] | 100.0 [97.6 to 100.0]
  Additional Serotypes - Serotype 7F (n= 84,108,142) | 100.0 [95.7 to 100.0] | 100.0 [96.6 to 100.0] | 99.3 [96.1 to 100.0]
  Additional Serotypes - Serotype 19A (n=84,110,150 | 100.0 [95.7 to 100.0] | 100.0 [96.7 to 100.0] | 100.0 [97.6 to 100.0]

2. Secondary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions
Description: Local reactions were collected using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (>7.0 cm). Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC Group 1 - Dose 1: Participants 7 to less than (<) 12 months of age with 0 prior doses of Prevnar received a single intramuscular (IM) 0.5 milliliter (mL) doses of 13-valent pneumococcal conjugate vaccine (13vPnC)(infant series).
- 13vPnC Group 2 - Dose 1: Participants 12 to < 24 months of age with 0 prior doses of Prevnar received a single IM 0.5 mL doses of 13vPnC (infant series).
- 13vPnC Group 3 - Dose 1: Participants 24 to < 72 months of age with 0 prior doses of Prevnar received a single IM 0.5 mL dose of 13vPnC (infant series).
- 13vPnC Group 1 - Dose 2: Participants 7 to less than (<) 12 months of age received a second single intramuscular (IM) 0.5 milliliter (mL) doses of 13-valent pneumococcal conjugate vaccine (13vPnC) at least 28 days after the first (infant series).
- 13vPnC Group 2 - Dose 2: Participants 12 to < 24 months of age received a second single IM 0.5 mL doses of 13vPnC at least 56 days from the first (infant series).
- 13vPnC Group 1 - Dose 3: Participants received a third single IM 0.5 mL dose of 13vPnC at 12 to 16 months of age (toddler dose), at least 46 days after last infant dose.
Arm/Group | 13vPnC Group 1 - Dose 1 | 13vPnC Group 2 - Dose 1 | 13vPnC Group 3 - Dose 1 | 13vPnC Group 1 - Dose 2 | 13vPnC Group 2 - Dose 2 | 13vPnC Group 1 - Dose 3
Number analyzed (Participants) | 90 | 112 | 152 | 90 | 112 | 89
percentage of participants
  Tenderness - Any | 15.1 | 33.3 | 42.3 | 15.1 | 43.7 | 15.2
  Tenderness - Significant | 1.2 | 0.0 | 4.1 | 3.5 | 4.1 | 6.4
  Swelling - Any | 36.0 | 44.5 | 36.9 | 32.2 | 41.0 | 25.0
  Swelling - Mild | 32.6 | 36.7 | 28.2 | 28.7 | 36.2 | 20.5
  Swelling - Moderate | 11.6 | 24.8 | 20.3 | 14.0 | 12.1 | 11.3
  Swelling - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Redness - Any | 48.8 | 70.0 | 50.0 | 46.0 | 54.7 | 37.8
  Redness - Mild | 41.9 | 55.5 | 37.4 | 40.2 | 44.7 | 31.3
  Redness - Moderate | 16.3 | 38.2 | 25.7 | 9.3 | 25.5 | 12.5
  Redness - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

3. Secondary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events
Description: Systemic events (fever ≥ 37.5 degrees Celsius [C], fever ≥ 38 C but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C, decreased appetite, irritability, increased sleep, decreased sleep, hives, use of medication to treat symptoms, and use of medication to prevent symptoms) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all subjects who received at least 1 dose of vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Group 1 - Dose 1 | 13vPnC Group 2 - Dose 1 | 13vPnC Group 3 - Dose 1 | 13vPnC Group 1 - Dose 2 | 13vPnC Group 2 - Dose 2 | 13vPnC Group 1 - Dose 3
Number analyzed (Participants) | 90 | 112 | 152 | 90 | 112 | 89
percentage of participants
  Fever ≥38°C but ≤39°C | 3.4 | 3.7 | 0.7 | 8.1 | 5.1 | 5.1
  Fever >39°C but ≤40°C | 1.2 | 0.9 | 0.7 | 2.3 | 0.0 | 1.3
  Fever >40°C | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Decreased appetite | 19.5 | 22.2 | 16.3 | 17.2 | 25.5 | 17.5
  Irritability | 24.1 | 30.6 | 14.3 | 34.5 | 34.0 | 24.7
  Increased sleep | 9.2 | 13.0 | 11.6 | 9.3 | 10.1 | 2.6
  Decreased sleep | 24.1 | 19.4 | 6.8 | 18.4 | 20.4 | 15.0
  Use of antipyretic medication to treat symptoms | 9.2 | 10.1 | 2.7 | 9.3 | 13.3 | 7.6
  Use of antipyretic medication to prevent symptoms | 8.0 | 13.8 | 4.8 | 4.7 | 14.3 | 5.1

4. Primary Outcome: Geometric Mean Antibody Concentration (GMC) After Vaccination in 13vPnC Groups
Description: GMC as measured by enzyme-linked immunosorbent assay (ELISA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: as for outcome 1
Population: The evaluable immunogenicity (per protocol) population was the primary analysis population consisting of eligible subjects who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC 7 to <12 Months of Age | 13vPnC 12 to <24 Months of Age | 13vPnC 24 to < 72 Months of Age
Number analyzed (Participants) | 84 | 110 | 152
μg/mL
  Common Serotypes - Serotype 4 | 3.63 [3.11 to 4.23] | 4.28 [3.78 to 4.86] | 3.37 [2.95 to 3.85]
  Common Serotypes - Serotype 6B | 4.77 [3.90 to 5.84] | 3.38 [2.81 to 4.06] | 3.41 [2.80 to 4.16]
  Common Serotypes - Serotype 9V | 2.56 [2.21 to 2.96] | 3.08 [2.69 to 3.53] | 2.67 [2.32 to 3.07]
  Common Serotypes - Serotype 14 | 8.04 [6.95 to 9.30] | 6.45 [5.48 to 7.59] | 2.24 [1.71 to 2.93]
  Common Serotypes - Serotype 18C | 2.77 [2.39 to 3.23] | 3.71 [3.29 to 4.19] | 2.56 [2.17 to 3.03]
  Common Serotypes - Serotype 19F | 2.88 [2.35 to 3.54] | 3.07 [2.68 to 3.51] | 2.53 [2.14 to 2.99]
  Common Serotypes - Serotype 23F | 2.16 [1.82 to 2.55] | 1.98 [1.64 to 2.39] | 1.55 [1.31 to 1.85]
  Additional Serotypes - Serotype 1 | 2.88 [2.44 to 3.39] | 2.74 [2.37 to 3.16] | 1.78 [1.52 to 2.08]
  Additional Serotypes - Serotype 3 | 1.94 [1.68 to 2.24] | 1.86 [1.60 to 2.15] | 1.42 [1.23 to 1.64]
  Additional Serotypes - Serotype 5 | 2.85 [2.34 to 3.46] | 2.16 [1.89 to 2.47] | 2.33 [2.05 to 2.64]
  Additional Serotypes - Serotype 6A | 3.72 [3.12 to 4.45] | 2.62 [2.25 to 3.06] | 2.96 [2.52 to 3.47]
  Additional Serotypes - Serotype 7F | 5.30 [4.54 to 6.18] | 5.99 [5.40 to 6.65] | 4.92 [4.26 to 5.68]
  Additional Serotypes - Serotype 19A | 4.77 [4.28 to 5.33] | 4.94 [4.31 to 5.65] | 6.03 [5.22 to 6.97]

ADVERSE EVENTS:
Arm/Group | 13vPnC 7 to <12 Months of Age | 13vPnC 12 to <24 Months of Age | 13vPnC 24 to < 72 Months of Age
Serious Adverse Events (participants affected / at risk) | 5/90 | 2/112 | 2/152
Other Adverse Events (participants affected / at risk) | 55/90 | 77/112 | 74/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC 7 to <12 Months of Age (N=90) | 13vPnC 12 to <24 Months of Age (N=112) | 13vPnC 24 to < 72 Months of Age (N=152)
Diarrhoea (General disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Exanthema subitum (Infections and infestations) | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC 7 to <12 Months of Age (N=90) | 13vPnC 12 to <24 Months of Age (N=112) | 13vPnC 24 to < 72 Months of Age (N=152)
Chalazion (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 8 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 1
Teething (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 2 | 1
Injection site nodule (General disorders) | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Allergy to animal (Immune system disorders) | 0 | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 12 | 13 | 5
Nasopharyngitis (Infections and infestations) | 11 | 12 | 5
Upper respiratory tract infection (Infections and infestations) | 8 | 16 | 4
Bronchitis (Infections and infestations) | 6 | 9 | 1
Respiratory tract infection (Infections and infestations) | 6 | 0 | 1
Rhinitis (Infections and infestations) | 6 | 9 | 4
Exanthema subitum (Infections and infestations) | 4 | 2 | 0
Viral infection (Infections and infestations) | 4 | 2 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 4 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 4 | 1
Varicella (Infections and infestations) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Urological examination abnormal (Investigations) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tenderness (any) (Skin and subcutaneous tissue disorders) | 13/86 | 36/108 | 63/149 — Infant Series Dose 1; Tenderness (any)=present at site of vaccination.
Tenderness (any) (Skin and subcutaneous tissue disorders) | 13/86 | 45/103 | 0/0 — Infant Series Dose 2; Tenderness (any)
Tenderness (any) (Skin and subcutaneous tissue disorders) | 12/79 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (any)
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 1/86 | 0/108 | 6/147 — Infant Series Dose 1; Tenderness (significant)=present and interfered with limb movement.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 3/86 | 4/98 | 0/0 — Infant Series Dose 2; Tenderness (significant)
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 5/78 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)
Induration (Any) (Skin and subcutaneous tissue disorders) | 31/86 | 49/110 | 55/149 — Infant Series Dose 1; Induration (any)=present at site of vaccination.
Induration (Any) (Skin and subcutaneous tissue disorders) | 28/87 | 43/105 | 0/0 — Infant Series Dose 2; Induration (Any)
Induration (Any) (Skin and subcutaneous tissue disorders) | 20/80 | 0/0 | 0/0 — Infant Series Dose 3; Induration (Any)
Induration (mild) (Skin and subcutaneous tissue disorders) | 28/86 | 40/109 | 42/149 — Infant Series Dose 1; Induration (mild)=0.5 centimeters (cm) to 2.0 cm.
Induration (mild) (Skin and subcutaneous tissue disorders) | 25/87 | 38/105 | 0/0 — Infant Series Dose 2; Induration (mild)
Induration (mild) (Skin and subcutaneous tissue disorders) | 16/78 | 0/0 | 0/0 — Infant Series Dose 3; Induration (mild)
Induration (moderate) (Skin and subcutaneous tissue disorders) | 10/86 | 27/109 | 30/148 — Infant Series Dose 1; Induration (moderate)=2.5 cm to 7.0 cm.
Induration (moderate) (Skin and subcutaneous tissue disorders) | 12/86 | 12/99 | 0/0 — Infant Series Dose 2; Induration (moderate)
Induration (moderate) (Skin and subcutaneous tissue disorders) | 9/80 | 0/0 | 0/0 — Infant Series Dose 3; Induration (moderate)
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/86 | 0/108 | 0/147 — Infant Series Dose 1; Induration (severe) >7.0 cm.
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/86 | 0/98 | 0/0 — Infant Series Dose 2; Induration (severe)
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/78 | 0/0 | 0/0 — Infant Series Dose 3; Induration (severe)
Erythema (any) (Skin and subcutaneous tissue disorders) | 42/86 | 77/110 | 74/148 — Infant Series Dose 1; Erythema (any)=present at site of vaccination.
Erythema (any) (Skin and subcutaneous tissue disorders) | 40/87 | 58/106 | 0/0 — Infant Series Dose 2; Erythema (any)
Erythema (any) (Skin and subcutaneous tissue disorders) | 31/82 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (any)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 36/86 | 61/110 | 55/147 — Infant Series Dose 1; Erythema (mild)=0.5 centimeters (cm) to 2.0 cm.
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 35/87 | 46/103 | 0/0 — Infant Series Dose 2; Erythema (Mild)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 25/80 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Mild)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 14/86 | 42/110 | 38/148 — Infant Series Dose 1; Erythema(moderate)=2.5 cm to 7.0 cm.
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 8/86 | 26/102 | 0/0 — Infant Series Dose 2; Erythema (Moderate)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 10/80 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Moderate)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/86 | 0/108 | 0/147 — Infant Series Dose 1; Erythema (severe) >7.0 cm.
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/86 | 0/98 | 0/0 — Infant Series Dose 2; Erythema (Severe)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/78 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Severe)
Fever ≥38°C but ≤39°C (General disorders) | 3/87 | 4/108 | 1/147 — Infant Series Dose 1; Fever ≥38°C but ≤39°C
Fever ≥38°C but ≤39°C (General disorders) | 7/86 | 5/98 | 0/0 — Infant Series Dose 2; Fever ≥38°C but ≤39°C
Fever ≥38°C but ≤39°C (General disorders) | 4/78 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥38°C but ≤39°C
Fever >39°C but ≤40°C (General disorders) | 1/86 | 1/108 | 1/147 — Infant Series Dose 1; Fever >39°C but ≤40°C
Fever >39°C but ≤40°C (General disorders) | 2/86 | 0/98 | 0/0 — Infant Series Dose 2; Fever >39°C but ≤40°C
Fever >39°C but ≤40°C (General disorders) | 1/79 | 0/0 | 0/0 — Infant Series Dose 3; Fever >39°C but ≤40°C
Fever >40°C (General disorders) | 0/86 | 0/108 | 0/147 — Infant Series Dose 1; Fever >40°C
Fever >40°C (General disorders) | 0/86 | 0/98 | 0/0 — Infant Series Dose 2; Fever >40°C
Fever >40°C (General disorders) | 0/78 | 0/0 | 0/0 — Infant Series Dose 3; Fever >40°C
Decreased appetite (General disorders) | 17/87 | 24/108 | 24/147 — Infant Series Dose 1; Decreased appetite
Decreased appetite (General disorders) | 15/87 | 25/98 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 14/80 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 21/87 | 33/108 | 21/147 — Infant Series Dose 1; Irritability
Irritability (General disorders) | 30/87 | 34/100 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 20/81 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 8/87 | 14/108 | 17/147 — Infant Series Dose 1; Increased sleep
Increased sleep (General disorders) | 8/86 | 10/99 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 2/78 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 21/87 | 21/108 | 10/148 — Infant Series Dose 1; Decreased sleep
Decreased sleep (General disorders) | 16/87 | 20/98 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 12/80 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.